CLINICAL TRIAL: NCT03502083
Title: Vasodilatory Effect of GLP-1
Brief Title: Human Vasodilatory Effect of GLP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14/EE/0018
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Coronary Stenosis; Type2 Diabetes; Angina, Stable
MeSH Terms: conditions — Coronary Stenosis; Angina, Stable | interventions — glucagon-like peptide 1 (7-36)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: GLP-1 (7-36)Amide — IV infusion

SUMMARY:
Comprehensive assessment of human vasodilatory effect of GLP-1 in forearm and coronary arteries

ELIGIBILITY:
Inclusion Criteria:

* Waiting list for elective PCI to LAD Able to give informed consent Over 18

Exclusion Criteria:

* GLP-1 based therapy Insulin Calcium channel blockers Nicorandil Nitrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Change in IMR (index of microcirculatory resistance) with GLP-1 compared with baseline | Change from baseline
  Change in coronary microcirculatory resistance from baseline
Forearm bloodflow ratio with GLP-1 | Change from baseline
  Peripheral vasodilatory response of GLP-1

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aetesam-Ur-Rahman M, Zhao TX, Paques K, Oliveira J, Khialani B, Kyranis S, Braganza DM, Clarke SC, Bennett MR, West NEJ, Hoole SP. Coronary Flow Variations Following Percutaneous Coronary Intervention Affect Diastolic Nonhyperemic Pressure Ratios More Than the Whole Cycle Ratios. J Am Heart Assoc. 2022 May 3;11(9):e023554. doi: 10.1161/JAHA.121.023554. Epub 2022 Apr 26. PMID 35470686
- [Derived] Aetesam-Ur-Rahman M, Giblett JP, Khialani B, Kyranis S, Clarke SJ, Zhao TX, Braganza DM, Clarke SC, West NEJ, Bennett MR, Hoole SP. GLP-1 vasodilatation in humans with coronary artery disease is not adenosine mediated. BMC Cardiovasc Disord. 2021 May 1;21(1):223. doi: 10.1186/s12872-021-02030-5. PMID 33932990